CLINICAL TRIAL: NCT06899542
Title: HEPATITIS C SCREENING in ADULTS with RISK FACTORS in FIVE CITIES of COLOMBIA'S CARIBBEAN COAST
Brief Title: HEPATITIS C SCREENING in ADULTS with RISK FACTORS in FIVE CITIES of COLOMBIA'S CARIBBEAN COAST (FIVE-CC)
Acronym: FIVE-CC
Status: Not yet recruiting | Type: Observational
Sponsor: Diana Rocio Chavez Bejarano (Other)
Responsible Party: Sponsor-Investigator, Diana Rocio Chavez Bejarano, DR., Asociación Colombiana de Hepatología
Organization: Asociación Colombiana de Hepatología (Other)
Other Study IDs: CO-US-987-7107
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C, general population.
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Hepatitis C virus (HCV) infection is a significant cause of chronic hepatitis, cirrhosis, and liver cancer (1). The risk of developing cirrhosis in people with chronic HCV infection ranges between 15% and 30% over a period of 20 years (2).

In 2016, the World Health Organization (WHO) defined the global strategy for eliminating viral hepatitis (Hepatitis C and Hepatitis B). The goals for hepatitis C include a 90% reduction in new cases of infection and a 65% reduction in mortality (3). To achieve this target by 2030, 90% of people living with hepatitis C need to be diagnosed, and 80% of those individuals must receive treatment, along with reducing the incidence of HCV in high-risk groups (4, 5).

According to 2019 data from the World Health Organization (WHO), 58 million people are living with chronic hepatitis C infection, (2).

Based on information from Colombia's High-Cost Account (CAC), between January 1 and December 31, 2021, 962 people with the infection were identified in Colombia (6). The CAC report for 2021 indicates that the prevalence of chronic HCV was 442, 173, 102, 089, and 25 cases per 100,000 inhabitants for Barranquilla, Soledad, Montería, Cartagena, and Santa Marta, respectively (7). The most common modes of transmission were sexual (72.1%) and parenteral/percutaneous (11.8% of cases) (8).

According to data published by the Polaris Observatory as of 2021, the prevalence in Colombia was estimated at 0.67% (320,000 cases), According to their projections, Colombia is expected to achieve the WHO targets by 2051 under current conditions (9).

Fewer than half of Latin American countries have conducted prevalence studies for HCV, and most of those studies have poor design quality. When extrapolating data from countries with records, the estimated HCV prevalence rate in Latin America is less than 1%. According to the Polaris Observatory's 2019 epidemiological data,only Brazil treated enough patients to achieve a net annual cure rate above 1% of those infected (10).

This study seeks to evaluate the prevalence of hepatitis C through rapid antibody testing and subsequent confirmatory quantitative viral load in the adult population with risk factors in five cities of the Colombian Caribbean coast: Barranquilla, Soledad, Montería, Cartagena, and Santa Marta.

DETAILED DESCRIPTION:
As of 2017, according to a WHO report, only 20% of people with HCV worldwide had been diagnosed (18). Micro- elimination strategies targeting small populations, rather than nationwide elimination programs, have been shown to improve diagnosis and treatment rates, yielding significant benefits for expanding the HCV care cascade and achieving WHO goals (14).

In the general population and the most affected populations, HCV screening recommendations from countries like Spain, the United Kingdom, Germany, France, Ireland, Canada, and Australia include population and opportunistic screening. This involves HCV screening in people exposed to risk factors such as intravenous or inhaled drug use, high-risk sexual behavior, HIV/HBV coinfection, aesthetic procedures involving sharp instruments without proper safety precautions, and imprisonment (17). Anyone who received blood transfusions before serological testing of blood donors for HCV, underwent medical or dental procedures in healthcare settings with substandard infection control practices, is also included.

Risk-based screening recommendations, as opposed to population screening, focus efforts and resources, ensuring equity in the design, implementation, and evaluation of HCV screening programs. These allow for addressing access barriers in each context (17). Targeted screening would identify a high number of infected individuals due to the higher infection rate related to risk factors, while simultaneously reducing viral transmission by eliminating HCV from individuals at higher risk of spreading the infection (20).

The study conducted by Rosato et al. (2022) highlight the need to increase awareness among general practitioners and other healthcare specialists who treat patients with different comorbidities to address HCV disease control. This is important as HCV eradication has been shown to significantly improve not only liver disease outcomes but also various comorbidities such as cryoglobulinemic vasculitis, diabetes, cardiovascular, and kidney diseases, etc. (21).

Monitoring the care cascade (CoC) is an essential component of the global response to the hepatitis C virus (HCV) epidemic. The findings allow healthcare decision-makers to determine where the most significant gaps in testing, care linkage, and treatment exist among people with chronic HCV infection (22).

Micro-elimination strategies in populations at high risk of transmitting HCV may contribute to the concept of "treatment as prevention." This concept involves successfully treating an HCV-infected individual who is at risk of transmitting the virus to others, thereby eliminating the possibility of further transmission, achieving "prevention." Due to its potential to prevent additional infections, many of which would incur high costs for treating end-stage liver disease, this approach could be highly cost-effective in the long term (18).

Targeting those at greatest risk of contracting the disease can generate broader community benefits and long-term cost-effectiveness. Supporting this approach to HCV eradication, model studies conducted by Martin and colleagues (2011 and 2013) have indicated that chronic HCV prevalence could be reduced by treating individuals at risk of continuous HCV transmission (23).

Since 2017, Colombia's High-Cost Account (CAC) has monitored identified chronic hepatitis C cases in accordance with Resolution 1692 of 2017, which is part of the strategy for negotiating and centrally purchasing direct-acting antivirals (24).

The most frequently used treatment in 98.2% of cases in the 2019-2020-2021 cohorts was sofosbuvir/velpatasvir, achieving 98.7% effectiveness in 2021 (25).

However, efforts are needed to incentivize screening in people over 50 years old and according to risk exposure, as established by Resolution 3280 of 2018 (25).

3. Research Question What is the prevalence of HCV in populations with risk factors for hepatitis C infection, detected through rapid testing in five cities on the Caribbean coast of Colombia? 4. Objectives

General Objective:

Determine the prevalence of HCV in patients with HCV risk factors, detected through opportunistic screening in five cities on the Caribbean coast of Colombia.

Specific Objectives:

* Characterize the sociodemographic profile of the study population.
* Describe the epidemiological characteristics of patients with positive HCV antibodies.
* Determine the proportion of patients with positive HCV antibodies and positive (quantitative) viral load for HCV.
* Conduct an exploratory analysis of the association between positive cases and various HCV infection risk factors.

  5. Methodology

Study Type:

Descriptive, cross-sectional, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

Present at least one of the following risk factors for hepatitis C:

* People over 50 years old with or without risk factors.
* People aged 18 and under 50 years old with risk factors for hepatitis C:

Individuals who have undergone medical or dental interventions in healthcare settings, Individuals with tattoos, body piercings, or scarification, Individuals co-infected with HIV or hepatitis B, People who inject drugs, Individuals who have used intranasal drugs, Individuals currently or previously incarcerated, Anyone with abnormal liver tests or liver disease, Healthcare students, workers, or public safety personnel (e.g., prison officers or police) who have been exposed to blood at work through needle-stick injuries or sharp objects, Sex workers, Men who have sex with men, Users of port health services, Reinserted or reintegrated individuals, Anyone who has undergone hemodialysis, Individuals who received blood transfusions in Colombia before 1996, People with comorbidities potentially associated with HC: diabetes, ischemic heart disease, cryoglobulinemia, chronic kidney disease, Sjögren's syndrome, hypothyroidism, lichen planus, rheumatoid arthritis, HIV, non-Hodgkin's lymphoma, acute lymphoblastic leukemia, Waldenström's macroglobulinemia, Individuals previously treated for HCV with a sustained viral response, where reinfection is suspected (individuals who continue to engage in risk behaviors). Confirmation testing through HCV viral load (PCR HCV) will be considered for inclusion in the study.

- Agree to participate in the study by signing an informed consent form.

Exclusion Criteria:

* Have had hepatitis C within the last three months with a confirmed cure by viral load 12 weeks after treatment or are actively receiving treatment for HCV and do not continue to engage in risk behaviors for reinfection.
* Voluntarily and knowingly refuse to sign the informed consent form or are unable to provide consent due to any type of physical and/or mental disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All individuals over the age of 18 with HCV risk factors, including the general population and vulnerable populations at higher risk of chronic hepatitis C infection, recruited from healthcare institutions or during screening campaigns in various settings.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
hepatitis C viremic | 5months
  HCV RNA detectable by quantitative method.

CONTACTS AND LOCATIONS:
Overall Officials: JAVIER E HERNANDEZ-BLANCO, DR, Principal Investigator — Asociación Colombiana de Hepatología; ISMAEL YEPES, DR, Principal Investigator — Asociación Colombiana de Hepatología

IPD SHARING:
Plan to Share IPD: No
Not included in the approved protocol